CLINICAL TRIAL: NCT04936464
Title: Transcutaneous Tibial Nerve Stimulation for Urgency Urinary Incontinence: A Sham-Controlled Trial
Brief Title: Transcutaneous Tibial Nerve Stimulation for Urgency Urinary Incontinence
Acronym: TTeNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12791
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Urge Incontinence; Overactive Bladder
Keywords: tibial nerve stimulation; transcutaneous electrical nerve stimulation; overactive bladder; urgency urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): 30-minute treatments, twice weekly x12 weeks
  Interventions: Device: transcutaneous tibial nerve stimulation (TTNS)
- Sham Group (Sham Comparator): 30-minute treatments, twice weekly x12 weeks
  Interventions: Device: transcutaneous electrical stimulation (TENS)

INTERVENTIONS:
Device: transcutaneous tibial nerve stimulation (TTNS) — TTNS is a non-invasive, surface electrode therapeutic stimulation technique available for home administration that has been proposed as a treatment for overactive bladder.
  Arms: Intervention Group
Device: transcutaneous electrical stimulation (TENS) — The sham intervention is designed to appear almost identical to the TTNS intervention.
  Arms: Sham Group

SUMMARY:
This is a single-center, double-blinded, randomized controlled trial evaluating the efficacy of TTNS versus a sham intervention. Both interventions will be performed by participants in their homes after standardized instruction. The primary outcome is a comparison of the mean change in OAB-q scores before and after treatment between the intervention and control groups. Changes in the number of urgency incontinence episodes and an estimation of cost effectiveness will additionally be measured. Intention to treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 episodes urgency incontinence on 3-day voiding diary
* Duration of symptoms ≥ 3 months
* Off antimuscarinic or 3-adrenoreceptor agonist therapy for 2 weeks
* No known neurologic disease
* Ability to complete home sessions and clinic follow up
* Ability to complete voiding diaries
* Internet access and proficiency
* English or Spanish-speaking

Exclusion Criteria:

* Pregnant
* Known or suspected urinary retention
* Symptomatic urinary tract infection unresolved at the time of randomization
* Recurrent urinary tract infection (≥ 3/12 months)
* Bladder pain syndrome
* Known or suspected advanced (stage III or IV) pelvic organ prolapse
* Neurogenic bladder
* Current or prior bladder malignancy
* Current or previous use of bladder Botox injections, percutaneous tibial nerve stimulation, or sacral neuromodulation
* Pacemaker or other implantable device
* Disease affecting lower extremities
* Bilateral metallic lower limb implant
* Incarceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Trial is open to biologically female participants only as this is the target population of interest.
Enrollment: 99 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Questionnaire (OAB-q) | 12 weeks
  To evaluate the efficacy of a 12-week course of TTNS in reducing urgency urinary incontinence (UUI) symptom bother in the intervention versus sham group.

SECONDARY OUTCOMES:
Voiding diary | 12 weeks
  To evaluate the efficacy of a 12-week course of TTNS in reducing the frequency of UUI episodes in the intervention versus sham group.

OTHER OUTCOMES:
Incremental cost-effectiveness ratio (ICER) | 12 weeks
  To describe the cost effectiveness of a 12-week course of home-based TTNS therapy using an ICER calculated from the sum of direct medical and indirect non-medical costs relative to health-related quality of life, as measured by the European Quality of Life-5 Dimensions index.

CONTACTS AND LOCATIONS:
Overall Officials: Nemi M Shah, MD, Principal Investigator — University of California San Diego/Kaiser Permanente San Diego
Locations (1):
- Kaiser Permanente San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah NM, Lukacz ES, Ferrante KL, Menefee SA. Transcutaneous Tibial Nerve Stimulation for Urge Incontinence: A Randomized Clinical Trial. Urogynecology (Phila). 2025 Mar 1;31(3):225-233. doi: 10.1097/SPV.0000000000001616. Epub 2024 Dec 13. PMID 39621424